CLINICAL TRIAL: NCT06777082
Title: Ruolo Delle Alterazioni Della Proteina RPL8 Nel Carcinoma Ovarico Sieroso ad Alto Grado
Brief Title: Role of RPL8 Protein Alterations in High-grade Serous Ovarian Carcinoma
Acronym: OVCAR
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: OVCAR; RC-22000593 (Other Grant/Funding Number: Ministero della Salute, Italy)
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: High Grade Serous Ovarian Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — DNA from post operators tissue specimen will be extracted for RPL8 & MYC status evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background and rationale of the study:

From our preliminary analyses of a dataset on patients with high-grade serous ovarian carcinoma (HGSOC), available in the online database The Cancer Genome Atlas, we found that the gene encoding ribosomal protein L8 (RPL8) is amplified at a high frequency (~30%) in HGSOC. Moreover, its mRNA expression is positively correlated with its genetic amplification-an observation not previously reported or studied in the literature. RPL8 is a structural component of the large ribosomal subunit, which is involved in protein synthesis. Based on this, and our preliminary data, we hypothesize that RPL8 amplification may play a role in ovarian cancer development. Understanding the impact of RPL8 amplification in ovarian cancer could provide new insights into the biology of this poorly understood cancer.

Study objectives:

The main objective of this project is to determine whether RPL8 can be used as a biomarker both for risk assessment and for patient stratification in choosing the most appropriate therapeutic option. Specifically, we aim to study:

1. The relationship between the genetic status of RPL8 and clinical outcomes.
2. The contribution of RPL8 amplification to treatment response.

Type of human tissue under study:

The analyses will be conducted on tumor tissue samples obtained from ovarian cancer resections. Some samples have already been collected and stored at the IRCCS, while others are yet to be gathered.

Type of investigation:

* Expression analysis of RPL8, C-MYC, and related genes (RT-PCR, ddPCR, WB, IHC).
* Gene copy number analysis and mutation screening (ddPCR and similar molecular techniques).
* Analysis of possible associations between pathological data, follow-up data, and therapeutic response outcomes in patients.

Analysis methodology:

Data on the genetic status, expression, and subcellular localization of RPL8 and C-MYC will be correlated with categorical and continuous variables related to the patients' medical history and clinical status. Differences between categorical variables will be analyzed using analysis of variance (ANOVA), the Mann-Whitney test, or the Kruskal-Wallis test, depending on whether data distribution is normal or not (assessed via the Kolmogorov-Smirnov test). Correlations between continuous variables will be evaluated using Pearson or Spearman tests, again based on data distribution.

DETAILED DESCRIPTION:
Background and rationale of the study:

From our preliminary analyses of a dataset on patients with high-grade serous ovarian carcinoma (HGSOC), available in the online database The Cancer Genome Atlas, we found that the gene encoding ribosomal protein L8 (RPL8) is amplified at a high frequency (~30%) in HGSOC. Moreover, its mRNA expression is positively correlated with its genetic amplification-an observation not previously reported or studied in the literature. RPL8 is a structural component of the large ribosomal subunit, which is involved in protein synthesis. Based on this, and our preliminary data, we hypothesize that RPL8 amplification may play a role in ovarian cancer development. Understanding the impact of RPL8 amplification in ovarian cancer could provide new insights into the biology of this poorly understood cancer.

Study objectives:

The main objective of this project is to determine whether RPL8 can be used as a biomarker both for risk assessment and for patient stratification in choosing the most appropriate therapeutic option. Specifically, we aim to study:

1. The relationship between the genetic status of RPL8 and clinical outcomes.
2. The contribution of RPL8 amplification to treatment response.

Type of human tissue under study:

The analyses will be conducted on tumor tissue samples obtained from ovarian cancer resections. Some samples have already been collected and stored at the IRCCS, while others are yet to be gathered.

Type of investigation:

* Expression analysis of RPL8, C-MYC, and related genes (RT-PCR, ddPCR, WB, IHC).
* Gene copy number analysis and mutation screening (ddPCR and similar molecular techniques).
* Analysis of possible associations between pathological data, follow-up data, and therapeutic response outcomes in patients.

Analysis methodology:

Data on the genetic status, expression, and subcellular localization of RPL8 and C-MYC will be correlated with categorical and continuous variables related to the patients' medical history and clinical status. Differences between categorical variables will be analyzed using analysis of variance (ANOVA), the Mann-Whitney test, or the Kruskal-Wallis test, depending on whether data distribution is normal or not (assessed via the Kolmogorov-Smirnov test). Correlations between continuous variables will be evaluated using Pearson or Spearman tests, again based on data distribution.

General characteristics of the study population:

Inclusion criteria:

* Age ≥ 18 years.
* Diagnosis of high-grade (3 or 4) serous ovarian carcinoma, either at onset or recurrence.
* Signed informed consent to participate in the study.

Exclusion criteria:

* Ovarian tumors of histological types other than serous.
* Other primary tumor types.

Study Design retrospective (on archival material) + prospective

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Diagnosis of high-grade (3 or 4) serous ovarian carcinoma, either at onset or recurrence.
* Signed informed consent to participate in the study.

Exclusion Criteria:

* Ovarian tumors of histological types other than serous.
* Other primary tumor types.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women affected with high grade serous ovarian cancer matching the inclusion criteria
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
RPL8 status | 2 years after enrollment
  RPL8 gene copy number and expression

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Montanaro, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azianda Ospedaliero-Universitaria di Bologna, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No